CLINICAL TRIAL: NCT05500872
Title: Blood Flow Restriction and Cross-education Effect on Muscle Strength Recovery After ACL Reconstruction
Brief Title: Blood Flow Restriction After Anterior Cruciate Ligament Reconstruction (ACLR)
Acronym: ACLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyda SEVINC, Reasearch Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19118
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Anterior Cruciate Ligament Rupture; Quadriceps Muscle Atrophy
Keywords: Anterior cruciate ligament; Strength training; Atrophy; Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Atrophy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Our study was planned to be randomized controlled. Individuals will be stratified into 2 groups (Group I, Group II) based on the order of arrival using the Excel program. After the 4th postoperative week, cross-training will be applied to both groups for 8 weeks in addition to the rehabilitation program. In the study group, cross-education will be performed for 8 weeks with blood flow restriction in the unaffected extremity in the isokinetic system. In the control group, cross-education will be performed for 8 weeks without applying blood flow restriction in the isokinetic system. Before and after cross education, individuals; pain (rest, activity), leg circumference measurement, quadriceps and hamstring muscle strength (isokinetic dynamometer), quadriceps muscle thickness, cross-sectional area (ultrasound) and knee function (IKDC questionnaire, KOOS questionnaire, tampa questionnaire) will be evaluated.
Who Masked: Outcomes Assessor
Masking Description: The thickness and cross-sectional area of the quadriceps muscle (rectus femoris, vastus medialis obliques, vastus lateralis) will be measured by ultrasonography before and after each participant's training (4th week and 12th week after surgery). The person making these measurements will not know which group the participants belong to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR Group (Experimental): Cross-education will be performed for 8 weeks with blood flow restriction in the unaffected extremity in the isokinetic system.
  Interventions: Other: Cross-education and blood flow restriction training
- Control Group (Active Comparator): Cross-education will be performed for 8 weeks without applying blood flow restriction in the isokinetic system.
  Interventions: Other: Cross-education

INTERVENTIONS:
Other: Cross-education and blood flow restriction training — Cross-education (training of the non-surgical leg) will be given to the participants in addition to the standard rehabilitation program after surgery. This training will be applied with isokinetic system that can be used safely in the rehabilitation field. During this training, a cuff will be worn from the upper part of the thigh muscles, as in the blood pressure devices, which will slow down the blood flow in the leg. The participant will be cross-educated with the cuff inflated to a safe pressure range that will not cause discomfort. Participants will be included in the training for a total of 16 sessions, 2 days a week for 8 weeks. Each session, cross-education will be applied as 3 sets of 12 repetitions. Pain, muscle strength, muscle thickness, knee functions will be evaluated before and after the training.
  Arms: BFR Group
Other: Cross-education — Cross-education (training of the non-surgical leg) will be given to the participants in addition to the standard rehabilitation program after surgery. This training will be applied with isokinetic system that can be used safely in the rehabilitation field. Participants will be included in the training for a total of 16 sessions, 2 days a week for 8 weeks. Each session, cross-education will be applied as 3 sets of 12 repetitions. Pain, muscle strength, muscle thickness, knee functions will be evaluated before and after the training.
  Arms: Control Group

SUMMARY:
Muscle strength and muscle volume decrease rapidly with the immobilization process after sports-related injury and surgery. Depending on the decrease in muscle strength and muscle volume, functional performance also deteriorates, and this has been demonstrated by studies in the literature. Despite rehabilitation programs after anterior cruciate ligament surgery, muscle weakness persists for a long time and this affects knee functions. As a result, the time to return to sports is delayed or the activity level decreases. In recent studies, cross training is used to gain strength. Cross training is the increase in strength in the untrained leg after unilateral strengthening of the untrained leg. Another popular application for strength gain is exercise training with blood flow restriction. Blood flow restriction exercise training is an exercise protocol based on external pressure restriction of blood flow through the cuff from the proximal of the target muscle. It has been shown that this training prevents reduction of muscle volume in the early postoperative period and increases muscle strength. In the literature, cross-training and blood flow-restricted training are applied separately for muscle strength development after ACL reconstruction. However, no study investigating the effect of the combined application of these two approaches on muscle strength during ACL rehabilitation has been found. It is thought that with the combined application of these approaches, their effects on muscle strength development will increase, and accordingly, the functional results of individuals will be positively affected. The aim of the study is to determine the effect of cross training applied with and without blood flow restriction on muscle strength and function for 8 weeks starting from the 4th week after anterior cruciate ligament surgery. Participants will be included in the training for a total of 16 sessions, 2 days a week for 8 weeks. Pain, muscle strength, muscle thickness, knee functions will be evaluated before and after the training.

DETAILED DESCRIPTION:
It has been suggested that standard strengthening exercises applied during rehabilitation after ACL reconstruction may be insufficient in terms of recovery of quadriceps strength and muscle volume. This insufficiency increases the risk of injury if the person returns to sports. At the same time, weight-bearing exercises within a safe knee range of motion are more recommended for these patients, as resistance quadriceps strengthening in non-weight-bearing positions (knee extension) for early strength gain is thought to be detrimental to graft healing. However, such exercises may not be as adequate as weightless exercises to strengthen the quadriceps. At this point, cross-training can be a potential way to achieve strength gain. Cross-education is an increase in strength in the untrained limb after unilateral strengthening of the homologous contralateral limb. Although the exact mechanisms of cross-education have not yet been defined, the strength gains produced in the non-exercising extremity are thought to occur as a result of improvements in cortical and spinal neural activity. Another popular practice for muscle hypertrophy recently is low-intensity exercise with blood flow restriction, also known as KAATSU training or occlusion training. Blood flow restriction exercise training is an exercise protocol based on external pressure restriction of blood flow by means of an elastic bandage or cuff from the proximal of the target muscle. It is recommended that external pressure be applied sufficiently to restrict venous return but maintain arterial flow. The relative anaerobic environment created during these periods of venous occlusion causes various localized cellular and hormonal changes that stimulate muscle hypertrophy. It is suggested that the effects of exercise increase in this hypoxic environment, thus increasing muscle mass and strength. It is thought that with the combined application of these approaches, their effects on muscle strength development will increase, and accordingly, the functional results of individuals will be positively affected.

The sample size was calculated as 1Nm/kg difference in muscle strength with 80% power and 0.05 type I error. A total of 20 individuals were determined, with 10 volunteers in each group.

Demographic information (age, gender, body mass index, dominant side, affected side, history, time from injury to surgery, date of surgery) of all cases will be recorded. Primary and secondary outcome meausers will be evaluated before the training session.

Eccentric cross-education with the isokinetic system will be applied to the unaffected extremities of the patients in the intervention and control groups. Each isokinetic training session will include 3 sets of 12 repetitions at 10°- 90° flexion angles, 60°/s angular velocity. There will be 2 minutes rest between sets. Cross-education will be applied in the same way for both groups. In the intervention group, blood flow restriction (occlusion) will be applied at a safe pressure range specific to each patient by wearing a pneumatic tourniquet from the proximal thigh during cross-training for 8 weeks.

The data will be analyzed using per-protocol anaylses. IBM SPSS 21.0 will be conducted for statistical analysis. The normality of the distribution will be analyzed with the Shapiro-Wilk test. The independent samples T test will be used for the normal distribution variables in the comparisons between the groups, and the Mann-Whitney U test will be used for the within-group comparisons for the variables that do not fit the normal distribution. For in-group comparisons, the paired samples T test will be used for the variables conforming to the normal distribution, and the Wilcoxon test will be used for the variables not conforming to the normal distribution. Significance level was set at p < 0.05.

If a patient is excluded from the study before his/her last assessment was conduded his/her date will be labelled as missing data. After the per-protocol analyses, the missing data will be replaced using the regression method. After the missing data replacement, the intention-to-treat analyses will be conducted using all data (per-protocol and missing data).

ELIGIBILITY:
Inclusion Criteria:

* Undergone reconstruction surgery with hamstring tendon graft due to unilateral anterior cruciate ligament tear,
* Absence of any injury in the intact extremity for at least 6 months
* Being recreationally active

Exclusion Criteria:

* Systemic or neurological problems
* History of deep vein thrombosis, peripheral vascular diseases
* Hypertension, cardiovascular diseases, neurological diseases, systemic inflammation, obesity, diabetes, atherosclerosis, advanced age)
* Active infection
* Having cancer
* Being pregnant
* Presence of posterior cruciate ligament tear in addition to the ACL
* Third degree tear in the lateral and medial collateral ligaments and and prominent articular cartilage lesion in addition to the ACL

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Muscle Strength at 12th week | 4th and 12th week after surgery
  Isometric muscle strength will be evaluated with isokinetic system. A 5-minute warm-up will be done before the test. After warming up, 5 repetitive hamstring stretching exercises will be performed on both extremities. The patients will then be seated on the isokinetic dynamometer seat with the trunk upright and the hips flexed to 90°, and the person will be positioned. The tests will be performed first on the unaffected side for each patient. Before starting the test, the test procedure will be explained to the patients in detail and the tests will be practiced once. For the quadriceps isometric muscle test, the patient will be asked to push the leg upwards with maximum force for 5 seconds. For the hamstring isometric muscle test, he will be asked to pull the leg down with maximum force. he test will be performed with three repetitions for each muscle and 2 minutes of rest will be given between repetitions to reduce the effect of fatigue. The results will be recorded in Nm/kg.

SECONDARY OUTCOMES:
Change from Baseline Muscle Thickness at 12th week | 4th and 12th week after surgery
  Ultrasound thickness (mm) and cross-sectional area (cm2) measurements of the quadriceps muscle will be used as primary outcome measure. Thickness measurement will be made on 3 parts of the quadriceps muscle (rectus femoris, vastus medialis oblique, vastus lateralis) using a B-mode ultrasound device (Siemens Medical Solution, Mountain View, CA, USA) and a Siemens 9L4 (4-9 MHz) linear probe. All measurements will be made at 25°C room temperature, in a darkened room, and by the same blinded radiologist who is unaware of the groups. Individuals will lie in the supine position during the measurement.
Change from Baseline Knee Function at 12th week | 4th and 12th week after surgery
  IKDC (International knee documentation committee) questionnaire will be used to evaluate the knee functions of the patients. The results will be recorded as scores.
Change from Baseline Knee Function at 12th week | 4th and 12th week after surgery
  KOOS (knee injury and osteoarthritis outcome score) questionnaire will be used to evaluate the knee functions of the patients. The results will be recorded as scores.
Change from Baseline Knee Function at 12th week | 4th and 12th week after surgery
  Tampa questionnaire will be used to evaluate the knee functions of the patients. The results will be recorded as scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided